CLINICAL TRIAL: NCT00002229
Title: A Phase IV, Non-Comparative Study to Evaluate FORTOVASE (Saquinavir) Soft Gel Capsule (SGC) TID Regimen in Combination With Two NRTI's in HIV-1 Infected Women and Men
Brief Title: Safety and Effectiveness of Adding Saquinavir (FORTOVASE) in Soft Gel Capsule Form to an Anti-HIV Drug Combination in HIV-Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 229Q; NR15750
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-12

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Dosage Forms; Saquinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Saquinavir

INTERVENTIONS:
Drug: Saquinavir

SUMMARY:
The purpose of this study is to see if it is safe and effective to give saquinavir (as a soft gel capsule taken by mouth) along with 2 other anti-HIV drugs to HIV-infected patients.

DETAILED DESCRIPTION:
Prior to initiation of study treatment all patients are screened and baseline lab values are taken. Patients then receive the study treatment, FORTOVASE, two times a day plus 2 new NRTI's. Assessments will be performed at specified intervals throughout the duration of treatment.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have an HIV count of 5,000 copies/ml or more.
* Have a CD4 count of 100 cells/mm3 or more.
* Meet specific requirements if you have ever taken NRTIs.
* Are 16 - 64 years old (need consent if under 18).
* Agree to use effective methods of birth control during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have taken non-nucleoside reverse transcriptase inhibitors (NNRTIs) or protease inhibitors (PIs) for more than 2 weeks.
* Have taken all the available NRTIs.
* Have certain serious medical conditions, including severe liver disease or active opportunistic (AIDS-related) infection.
* Have a history of weight loss, muscle pain, and loss of appetite.
* Have taken certain medications, including anti-HIV drugs other than those required by this study.
* Are pregnant or breast-feeding.
* Abuse alcohol or drugs.
* Are unable to complete the study for any reason.

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80

CONTACTS AND LOCATIONS:
Overall Officials: S Palleja, Study Chair; C Karol, Study Chair
Locations (22):
- United States (20):
  - ASC Inc, Hobson City, Alabama
  - Dean Martin, Phoenix, Arizona
  - Wilbert Jordan, Paramount, California
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - Duval County Health Department, Jacksonville, Florida
  - Ctr for Quality Care, Tampa, Florida
  - NTouch Research Corp, Decatur, Georgia
  - Univ of Illinois Hosp at Chicago, Chicago, Illinois
  - Univ of Kentucky, Lexington, Kentucky
  - C100 HIV Outpatient Program, New Orleans, Louisiana
  - NJ CRI, Newark, New Jersey
  - UMDNJ / Dept of Ob/Gyn, Newark, New Jersey
  - SUNY Health Sciences Ctr, Brooklyn, New York
  - Brookdale Univ Med Ctr, Brooklyn, New York
  - Mt Vernon Hosp, Mount Vernon, New York
  - Mount Sinai Med Ctr, New York, New York
  - Harlem Hosp Infectious Disease, New York, New York
  - Mem Hosp of Rhode Island, Pawtucket, Rhode Island
  - Diversified Med Practices, PA, Houston, Texas
  - Univ of Virginia Health Sciences Ctr, Charlottesville, Virginia
- Univ of British Columbia Oak Tree Clinic, Vancouver, British Columbia, Canada
- Programe DeSIDA De San Juan, Santurce, Puerto Rico